CLINICAL TRIAL: NCT01282255
Title: A Randomised, Double Blind, Placebo-controlled, Multiple Dose Trial of Anti-IL-20 (109-0012) in Subjects With Rheumatoid Arthritis
Brief Title: Efficacy of NNC109-0012 in Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8226-3875; U1111-1117-1136 (Other: WHO); 2010-021283-14 (EudraCT Number)
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: NNC109-0012
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC109-0012 — The subjects will receive 12 weekly doses of 3 mg/kg of NNC109-0012 administered subcutaneously (under the skin)
  Arms: A
Drug: placebo — The subjects will receive 12 weekly doses of 3 mg/kg of Placebo administered subcutaneously (under the skin)
  Arms: B

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the change in disease activity following 12 weekly s.c. (under the skin) doses of NNC109-0012 compared to placebo in subjects with active Rheumatoid Arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Czech Republic: Age between 18 - 65 years (both inclusive)
* A diagnosis of RA made at least 3 months prior to trial start
* Active RA
* Methotrexate treatment (between 7.5 mg and 25 mg/week, both inclusive) for at least 12 weeks with a stable dose for at least 4 weeks prior to trial start
* Female subjects must be willing to avoid pregnancy and breast feeding throughout this trial at least until 15 weeks following the last dose of trial medication
* Male subjects with partners of childbearing potential must be willing to use a highly effective contraception throughout trial incl. a 15 week follow up periode

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Body Mass Index (BMI) lower than 18.5 or higher than 35.0 kg/m^2
* Subjects with chronic inflammatory autoimmune disease other than RA (except secondary Sjögren's syndrome or stable hypothyroidism)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in DAS28-CRP (disease activity score 28 calculated with C-reactive protein value) | week 0, week 12

SECONDARY OUTCOMES:
Terminal serum half-life (t½) | end of treatment period
Serum levels of NNC109-0012 | end of treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (27):
- Czechia (4):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Prague
  - Novo Nordisk Investigational Site, Uherské Hradiště
  - Novo Nordisk Investigational Site, Zlín
- Germany (3):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Würzburg
- Novo Nordisk Investigational Site, Pavia, Italy
- Poland (7):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Bydgoszcz
  - Novo Nordisk Investigational Site, Bytom
  - Novo Nordisk Investigational Site, Elblag
  - Novo Nordisk Investigational Site, Gmina Końskie
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Żyrardów
- Novo Nordisk Investigational Site, Lisbon, Portugal
- Romania (4):
  - Novo Nordisk Investigational Site, Cluj-Napoca, Cluj
  - Novo Nordisk Investigational Site, Târgovişte, Dâmbovița County
  - Novo Nordisk Investigational Site, Ploieşti, Prahova
  - Novo Nordisk Investigational Site, Brăila
- Spain (4):
  - Novo Nordisk Investigational Site, A Coruña
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Seville
- United Kingdom (3):
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, Norwich

REFERENCES:
- [Result] Lundblad MS, Overgaard RV, Gothberg M, Fjording MS, Watson E. Clinical pharmacokinetics of the anti-interleukin-20 monoclonal antibody NNC0109-0012 in healthy volunteers and patients with psoriasis or rheumatoid arthritis. Adv Ther. 2015 Mar;32(3):228-38. doi: 10.1007/s12325-015-0191-7. Epub 2015 Mar 7. PMID 25749867
- [Result] Senolt L, Leszczynski P, Dokoupilova E, Gothberg M, Valencia X, Hansen BB, Canete JD. Efficacy and Safety of Anti-Interleukin-20 Monoclonal Antibody in Patients With Rheumatoid Arthritis: A Randomized Phase IIa Trial. Arthritis Rheumatol. 2015 Jun;67(6):1438-48. doi: 10.1002/art.39083. PMID 25707477
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com